CLINICAL TRIAL: NCT04917445
Title: A Comparison of the SPIKES Protocol for Delivering Bad News to the Current Standard of Care in the in Vitro Fertilization Population
Brief Title: The Impact of the SPIKES Protocol With IVF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston IVF (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Alice Domar, Executive Director of Domar Center for Mind Body Health, Boston IVF
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BN2021
Record Dates: First submitted 2021-05-26; First posted 2021-06-08 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Infertility
Keywords: infertility; IVF; Spikes protocol
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIKES Protocol Compassionate Call (Experimental): Nurses trained to contact IVF patients with negative pregnancy test results who were trained on the SPIKES-focused bad news delivery script.
  Interventions: Behavioral: Spikes-focused bad news protocol
- Control: Standard of Care Call (No Intervention): Nurses who will continue to deliver bad news as they have been in the past without a script.

INTERVENTIONS:
Behavioral: Spikes-focused bad news protocol — Nurses trained to deliver bad news to IVF patients based on the Spikes-protocol for compassionately delivering bad news to patients.
  Arms: SPIKES Protocol Compassionate Call

SUMMARY:
The purpose of this study is to determine if the utilization of the SPIKES protocol for delivering bad news is perceived to be more compassionate and effective than the current standard of care for IVF patients receiving negative pregnancy test results.

DETAILED DESCRIPTION:
Presently, nurses at Boston IVF (BIVF) and Weill Cornell Medical Center Division of Reproductive Medicine (Cornell) do not have a scripted method to deliver negative pregnancy tests to in Vitro Fertilization (IVF) patients. This study will invite clinic nurses to assist in the research protocol; half of the nurses will be randomized to be trained on a compassionate way to deliver bad news following the SPIKES protocol, while the other half will continue with the current standard of care of news delivery. The patients who receive the negative test phone calls from participating nurses will be surveyed to see if the method of which the news was delivered was scored as more compassionate, as well as if it was associated with reduced participants reported level of distress and depression.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age >18
* Underwent an embryo or blastocyst transfer using their own eggs at participating clinic
* Able to read and understand English
* Access to email
* Received a negative pregnancy test result phone call from a nurse involved in the research study

Exclusion Criteria:

* Partners of patients undergoing treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 136 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Assess if the SPIKES-based nursing script is associated with a difference in perceived nursing compassion | Within 48 hours of phone call
  We revised the Communicating Bad News questionnaire which follows the SPIKES protocol, published by Gonzales-Cabrera et al. Their questionnaire had 25 items, Internal consistency was 0.816. The content validity was established via the Kaiser-Meyer-Olkin test (KMO) with a score of 0.683 and the Bartlett test of sphericity was p<0.001. The principal component analysis supported a four dimension construct. There are 22 items rated 1, 2, 3 with a scoring range of 22-66. For the Compassion Assessment, there are 19 slots for the 5 categories so the scoring range is 5-95. The content validity was established via the Kaiser-Meyer-Olkin test (KMO) with a score of 0.683. and the Bartlett test of sphericity was p<0.001. The principal component analysis supported a four dimension construct. There are 22 items rated 1,2,3 so the scoring range is 22-66. For the Compassion Assessment, there are 19 slots for the 5 categories so the scoring range is 5-95.
Assess patient distress after receiving the negative pregnancy test phone call | Within 48 hours of phone call
  We will use 5-point Likert scales to assess patient distress after receiving the negative pregnancy test phone call. The Likert scale range is 1-5.
Assess patient depression after receiving the negative pregnancy test phone call | Within 48 hours of phone call
  We will use 5-point Likert scales to assess patient depression after receiving the negative pregnancy test phone call. The Likert scale range is 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Domar, PhD, Principal Investigator — Boston IVF
Locations (2):
- United States (2):
  - Boston IVF, Waltham, Massachusetts
  - Weill Cornell Medical Center Division of Reproductive Medicine, New York, New York

REFERENCES:
- [Derived] Domar AD, Korkidakis A, Bortoletto P, Gulrajani N, Khodakhah D, Rooney KL, Gompers A, Hacker MR, Grill E. The impact of an adapted SPIKES protocol vs routine care in the delivery of bad news to IVF patients: an exploratory pilot multicenter randomized controlled trial. J Assist Reprod Genet. 2024 Sep;41(9):2367-2377. doi: 10.1007/s10815-024-03198-3. Epub 2024 Jul 19. PMID 39026124